CLINICAL TRIAL: NCT03983616
Title: Surveillance of Invasive Pneumococcal Infections in Adults (Excluding Meningitis)
Acronym: SIIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Collaborators: INVS (Unknown); ORP (Unknown); CNRP (Unknown); SPILF (Unknown)
Responsible Party: Sponsor
Other Study IDs: SIIP
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Given the frequency and severity of invasive pneumococcal infections and questions about the place of VPC-13 in the prevention of pneumococcal infections in adults based on the presence of risk factors, current laboratory surveillance should be supplemented with data on the clinical features of adult invasive pneumococcal infections (IPI) cases. In particular it is necessary to collect for these cases, the clinical forms, the severity and the existence of risk factors and to make the link between these characteristics and those strains of pneumococci responsible for the IPI in particular, their serotype. The follow-up of the evolution of the cases according to the presence of risk factors, their clinical form and their serotype coverage (vaccine strain or not) must to guide recommendations for adult VPC-13 and to monitor the effects of VPC-13 vaccination recommendations. These effects are indirect, linked to the effect of vaccination of children with VPC-13 since 2010, which modifies the serotypes responsible for infections in vaccinated and unvaccinated patients, and the direct effects of possible use of the conjugate vaccine in adults (according to the recommendations that will be given by the Vaccination Technical Committee of the High Council of Public Health). The project is based on the existing network of 23 Regional Pneumococcal Observatories (ORP) located in metropolitan France and the network of infectious diseases by completing the microbiological collection of strains of pneumococci isolated from invasive infections in adults by a clinical collection in hospitals or voluntary clinics where the laboratory participates in the ORP. Given the establishment in 2012 of an adult bacterial meningitis observatory, to which the ORP are associated, this project does not include the surveillance of pneumococcal meningitis in adults.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old patients or older hospitalized with invasive pneumococcal infection confirmed by isolation of a strain from a usually sterile site: blood or pleural fluid

Exclusion Criteria:

* Pneumococcal meningitis identified by pneumococcal isolation or pneumococcal positive polymerase chain reaction (PCR) in cerebrospinal fluid

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults 18 years of age or older hospitalized for invasive pneumococcal disease in participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 1560 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of invasive pneumococcal infections | Day 0
  identify the frequency of invasive pneumococcal infections in function of the presence of risk factors

SECONDARY OUTCOMES:
Weight of invasive pneumococcal infections | Day 0
  measure the weight of invasive pneumococcal infections based on the presence of risk factors and immunization or not
Number of Invasive Pneumococcal Infections in Adults | Day 0
  monitor the epidemiology of Invasive Pneumococcal Infections in Adults according to strategies for the use of VPC-13 and VPS-23 vaccines in children and adults

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Virologie, Limoges, France